CLINICAL TRIAL: NCT03938025
Title: Impact of Resected Gastric Volume on Postoperative Weight Loss After Laparoscopic Sleeve Gastrectomy for Morbid Obesity
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Paolo Gentileschi, Bariatric Surgery Unit Chief, University of Rome Tor Vergata
Other Study IDs: Gastric Volume Sleeve
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Morbid Obesity
Keywords: Sleeve gastrectomy; Morbid obesity; Resected gastric volume
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Gastric volume resected in sleeve gastrectomy — Misure of resected gastric volume and outcome

SUMMARY:
Impact of resected gastric volume on postoperative weight loss after laparoscopic sleeve gastrectomy for morbid obesity. Observational study with a mathematical method to approximate the calculation of the resected gastric volume after a sleeve gastrectomy and see the outcome on weight loss.

ELIGIBILITY:
Inclusion Criteria:

* BMI over 60 kg/m2 in high-risk patients,
* BMI between 50 and 60 kg/m2 in nondiabetic patients,
* BMI between 40 and 50 kg/m2 in patients refusing a complex procedure like Roux-en-Y gastric bypass,
* patients with severe gastric inflammatory disease and H. pylori infection,
* patients with previous abdominal surgery involving the intestines, and young patients refusing gastric banding

Exclusion Criteria:

* severe and documented gastroesophageal reflux disease
* previous gastric surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: final group from which data have been considered 92 patients (47females and 45 males)
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
resected gastric volume in laparoscopic sleeve gastrectomy | 5 years
  Impact of resected gastric volume on postoperative weight loss after laparoscopic sleeve gastrectomy for morbid obesity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Ugo S, Bellato V, Bianciardi E, Gentileschi P. Impact of Resected Gastric Volume on Postoperative Weight Loss after Laparoscopic Sleeve Gastrectomy. Gastroenterol Res Pract. 2019 Dec 1;2019:3742075. doi: 10.1155/2019/3742075. eCollection 2019. PMID 31871448